CLINICAL TRIAL: NCT01243294
Title: Cross-over, Open Label Study Evaluating a New Ostomy Appliance With Regard to Leakage, Handling and Comfort
Brief Title: Study Evaluating a New Ostomy Appliance With Regard to Leakage, Handling and Comfort
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CP209OC
Record Dates: First submitted 2010-08-09; First posted 2010-11-18 (Estimated); Results first posted 2011-06-22 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SenSura (Active Comparator): CE marked and launched (The letters "CE" do not represent any specific words, though may have initially stood for "Communauté Européenne" ("European Community") or "Conformité Européenne" ("European Conformity"). By affixing the CE marking to a product, the manufacturer declares that it meets EU safety and health and environmental requirements.
  Interventions: Device: SS; Device: SenSura
- New ostomy appliance (SS) (Active Comparator): SS = New ostomy appliance. Due to company confidentiality the product is just called SS and this is not short for any other names.
  Interventions: Device: SS; Device: SenSura

INTERVENTIONS:
Device: SS — New ostomy appliance (SS) is tested in 10 ± 2 days and the degree of leakage under the baseplate is measured and compared to SenSura.
  Other Names: SenSura; New ostomy appliance
Device: SenSura — New ostomy appliance (SS) is tested in 10 ± 2 days and the degree of leakage under the baseplate is measured and compared to SenSura.
  Other Names: New ostomy appliance

SUMMARY:
The objective of this investigation is to evaluate leakage, handling and comfort of a new ostomy appliance compared to SenSura.

DETAILED DESCRIPTION:
Peristomal skin problems are reported to have a negative impact on the quality of life of people with a stoma and cause one third of all visits to a stoma care nurse. Stoma effluent in contact with the peristomal skin (leakage) appears to predispose patients to peristomal skin problems.

To protect the skin against effluent, the appliance used for collection of stoma effluent should completely cover the peristomal skin close to the stoma. Coloplast has developed a new ostomy appliance to improve the feeling of security and increase comfort by the appliance characteristics.

The objective of this investigation is to evaluate leakage, handling and comfort of a new ostomy appliance compared to SenSura.

The study is a randomised controlled cross-over intervention study, where all study participants will test two test products (new ostomy appliance and SenSura). Each test period will last 10 ± 2 days and the subjects will follow their usual wear and change pattern. The participants will visit the study investigator at study start and at cross-over. Evaluation of the test products will occur via questionnaires the subjects fill in at home.

50 healthy subjects with a colostomy will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Be at least 18 years of age and have full legal capacity
* Be able to handle the bags themselves (application, removal)
* Have a colostomy with a diameter less than 45 mm
* Have had a colostomy for at least 3 months
* Currently use a 1-piece flat ostomy appliance with closed bag
* is suitable for treatment with a standard adhesive, flat base plate (evaluated by nurse)
* Use minimum 1 product per day
* Be willing to test a new Coloplast one-piece custom cut ostomy appliance size midi or maxi for 10 days and SenSura (1- piece open ostomy bag custom cut ostomy appliance) size midi or maxi for 10 days
* Have the mental capacity to understand the study and questionnaires

Exclusion Criteria:

* Use irrigation during the study (flush the stoma with water).
* Currently suffering from peristomal skin problems (i.e. bleeding or red and broken skin)
* Currently receiving or have within the last 2 months received chemotherapy or radiation therapy
* Currently receive or have within the past three weeks been receiving steroid medication in the peristomal area.
* Are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pia Nordmand, MSc, Principal Investigator — Coloplast A/S
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from a user database in Denmark and through six hospital sites in France between august and november 2010
Pre-assignment Details: 56 subject where enrolled, however two subjects did not comply to the in- and exclusion criteria and was hence terminated before testing any devices
Groups:
- SenSura First, Then SS; SS First, Then SenSura: SS = new ostomy bag. SS used in this trial is a 1-piece closed ostomy product consisting of a base plate and a bag. The intended use is collecting output from a colostomy.
  SenSura used in this trial is a 1-piece closed ostomy product consisting of a base plate and a bag. The intended use is collecting output from a stoma (e.g. a ileostomy or a colostomy).
  Both SS and SenSura is changed 1 till 6 times a day, depending on when the bag is full, or if there is leakage.
  The difference between the two products is the adhesive on the base plate where SS have a softer adhesive than SenSura. It is this soft adhesive we wanted to test.
Period: First Intervention (10 Days +/- 2 Days)
Arm/Group | SenSura First, Then SS | SS First, Then SenSura
Started | 28 | 26
Completed | 28 | 26
Not Completed | 0 | 0
Period: Second Intervention (10 Days +/- 2 Days)
Arm/Group | SenSura First, Then SS | SS First, Then SenSura
Started | 28 | 26
Completed | 28 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive SS (new ostomy bag)first and SenSura first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 54
Age Continuous [Mean (Standard Deviation); unit: years] | 70.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 35
Region of Enrollment [Number; unit: participants]
  Denmark | 39
  France | 15

OUTCOME MEASURES:

1. Primary Outcome: Leakage (Percent of All Base Plates With Leakage)
Description: Leakage is evaluated after each change of base plate on a 4-point scale from no leakage, leakage on the base plate, leakage soiling clothe and sudden leakage - the 3 last mentioned are all defined as leakage. No leakage is the preferred end point
Time Frame: After each base plate change measured over a period of 10 +/- 2 days. Base plates are changed 1-6 times a day
Population: Intention to treat. As this is a cross-over investigation 26 started at SS and crossed over to SenSura, and 28 started at SenSura and crossed to SS leading to a total population of 54 evaluating each medical device
Measure: Number; unit: Percent of Base plates
Units Other Than Participants: Base plates
Groups:
- New Adhesive SS: SS = new adhesive. SS used in this trial is a 1-piece closed ostomy product consisting of a base plate and a bag. The intended use is collecting output from a colostomy.
  Both SS and SenSura is changed 1 till 6 times a day, depending on when the bag is full, or if there is leakage.
  The difference between the two products is the adhesive on the base plate where SS have a softer adhesive than SenSura. It is this soft adhesive we wanted to test.
- SenSura: CE marked and launched SenSura used in this trial is a 1-piece closed ostomy product consisting of a base plate and a bag. The intended use is collecting output from a stoma (e.g. a ileostomy or a colostomy).
  Both SS and SenSura is changed 1 till 6 times a day, depending on when the bag is full, or if there is leakage.
  The difference between the two products is the adhesive on the base plate where SS have a softer adhesive than SenSura. It is this soft adhesive we wanted to test.
Arm/Group | New Adhesive SS | SenSura
Number analyzed (Participants) | 54 | 54
Number analyzed (Base plates) | 975 | 1046
Percent of Base plates | 27 | 30

2. Secondary Outcome: Adverse Events
Description: Safety is evaluated by adverse events occuring continues while the subjects are testing the devices
Time Frame: During the investigation ~ 24 days per subject
Population: As this is a cross-over investigation 26 started at SS and crossed over to SenSura, and 28 started at SenSura and crossed to SS leading to a total population of 54 evaluating each medical device.
  Population is ITT
Measure: Number; unit: Adverse events
Arm/Group | New Adhesive SS | SenSura
Number analyzed (Participants) | 54 | 54
Adverse events | 1 | 2

3. Secondary Outcome: Security (Subjects Own Assessment)
Description: Results of participants who answered on own assessment of security on a 5 point scale ('very poor', 'poor', 'acceptable', 'good' and 'very good'). 'Good' and 'very good' are the preferred end points The 'very good' result are presented here.
  Unit of measure is: Percentage of participants answering 'very good'
Time Frame: After each test period, i.e. after 10 (±2) days with one test product and after 10 (±2) days with the other test product
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | New Adhesive SS | SenSura
Number analyzed (Participants) | 54 | 54
Percent of participants | 48 | 28

4. Secondary Outcome: Handling at Appliance (Subjects Own Assessment)
Description: Handling at appliance where evaluated by subjects own assessment on a 5 point scale from very difficult to very easy.
  Results of participants who answered on own feeling of handling at appliance on a 5 point scale (very difficult, difficult, acceptable, easy, very easy). Easy and very easy are the preferred end points and it is the these results that are presented here.
  Unit of measure is: Percentage of participants answering 'very easy' and 'easy'
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | New Adhesive SS | SenSura
Number analyzed (Participants) | 54 | 54
Percent of participants | 89 | 91

5. Secondary Outcome: Comfort (Subjects Own Assessment)
Description: Comfort where evaluated by subjects own assessment on a 5 point scale from very uncomfortable to very comfortable.
  Results of participants who answered on own assessment of comfort of wearing the product on a 5 point scale (very uncomfortable, uncomfortable, acceptable, comfortable, very comfortable). Comfortable and very comfortable are the preferred end points and it is these results that are presented here.
  Unit of measure is: Percentage of participants answering 'very comfortable' and 'comfortable'
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | New Adhesive SS | SenSura
Number analyzed (Participants) | 54 | 54
Percent of participants | 93 | 67

6. Secondary Outcome: Wear Time (Registered by Subject When Applying and Removing a Product)
Description: Wear time was calculated from the time the subjects applied their product (date, year, time) to the time they detached the product (date, year, time). Wear time was estimated in hours per subject per base plate and mean value was calculated.
Time Frame: After each base plate change measured over a period of 10 +/- 2 days. Base plates are changed 1-6 times a day
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Units Other Than Participants: Base plates
Arm/Group | New Adhesive SS | SenSura
Number analyzed (Participants) | 54 | 54
Number analyzed (Base plates) | 975 | 1046
Hours | 11.46 (7.07) | 11.41 (6.41)

ADVERSE EVENTS:
Time Frame: AE data where collected from inclusion to the two test periods where completed (~24 days)
Groups:
- SenSura: Base plates applied 1 till 6 times a day
- SS (New Ostomy Bag): Base plates applied 1 till 6 times a day SS = new ostomy bag
Arm/Group | SenSura | SS (New Ostomy Bag)
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 2/54 | 1/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SenSura (N=54) | SS (New Ostomy Bag) (N=54)
Redness and skin damage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rated as related to medical device. Moderate severity. Device used while experiencing adverse event: SenSura
Peripheral lesions from 5 cm (peripheral edges) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rated as related to medical device. Moderate severity. Device used while experiencing adverse event: SenSura
Redness on skin 0-2 cm from stoma edge (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Rated as related to medical device. Mild severity. Device used while experiencing adverse event: SS (new ostomy appliance)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes